CLINICAL TRIAL: NCT05091593
Title: A Hybrid Type I Randomized Effectiveness-Implementation Trial of Remote Treatment of Depression in Rural Community Cancer Centers
Brief Title: Intervention for Rural Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Steel, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY21060157
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Depression; Quality of Life; Social Support; Sleep; Stress
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Research Study Coordinators will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stepped collaborative care intervention (Experimental): The 'Stepped Collaborative Care Intervention' includes at least biweekly contact from a care coordinator by phone and face to face visits occurring approximately every 2 months, and 24 hour 7 day a week access to a website that was specifically designed during the pilot study for advanced cancer patients from socioeconomically disadvantaged backgrounds.
  Interventions: Behavioral: Stepped collaborative care intervention
- Enhanced Usual Care (Active Comparator): Patients randomized to the 'Enhanced Usual Care' arm receive their usual care from their medical team. However, if the patient scores in the clinical range on one or more of the three symptoms s/he will receive education about the symptom and be referred to the appropriate health care provider for further treatment in their community. The care coordinator will follow up with the patient after 3 weeks to assess barriers to treatment and assist further with accessing treatment if needed.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Stepped collaborative care intervention — Using website that was specifically designed for advanced cancer patient, collaborative with treatment from health professional.
  Other Names: Treatment
  Arms: Stepped collaborative care intervention
Behavioral: Enhanced Usual Care — Usual care from health providers
  Other Names: Control
  Arms: Enhanced Usual Care

SUMMARY:
In an effort to reduce rural-urban disparities and improve the quality of cancer care for these patients, the objectives of this study will be to: (1) adapt the intervention to maximize effectiveness for rural, low-income patients, (2) test the effectiveness of the adapted intervention, and (3) prepare for implementation of the intervention in rural, low-income communities.

DETAILED DESCRIPTION:
The purpose of the study is to reduce rural-urban disparities and improve the quality of cancer care for these patients:

(Aim 1): By using mixed methods, investigators will adapt the stepped collaborative care intervention to address the contextual needs of patients diagnosed with comorbid cancer and depression living in rural, low-income communities. Using face-to-face qualitative interviews with 30 patients diagnosed with cancer and quantitative data from our past trial, investigators will adapt the stepped collaborative care intervention for patients diagnosed with cancer from rural, low-income communities. For all quantitative data, the frequency distributions of study variables will be examined prior to statistical analyses to provide descriptive data and to identify departures from normality. If nonlinearity is detected, a transformation will be performed using the Box-Cox transformation, which finds the optimal relationship between variables. All measures have established reliability and validity similar to that from which the study sample will be drawn; however, the reliabilities of scales will be assessed using Cronbach's. Thorough exploratory data analyses will be performed to ascertain data characteristics and to screen for anomalies (i.e., outliers). The preliminary exploration of the data will be used to: (1) examine univariate and bivariate distributions; (2) identify any imbalances between treatment groups on baseline characteristics; (3) investigate the magnitude of the associations between the dependent variables and the potential covariates; (4) determine the internal consistency reliabilities of the measurement scales using Cronbach's alpha; and (5) verify the statistical assumptions of the planned primary analyses. If assumptions are violated, then alternative procedures such as data transformations or more robust statistical methods will be considered. Missing data will be examined using available data on subject characteristics. Logistic regression models will be created with SAS PROC LOGISTIC to compare the characteristics of subjects who remained in the study versus those who dropped out. If data are determined to be missing at random, likelihood estimation procedures available in SAS PROC MIXED will produce unbiased estimates and allow the retention of subjects with missing data on outcomes. If data are determined to be not missing at random, pattern mixture or selection modeling will be used to investigate attrition. If necessary, multiple imputation (SAS PROC MI) will be used to impute missing values for covariates.

(Aim 2): To test, in a randomized controlled trial, the adapted stepped collaborative care intervention for 242 patients diagnosed with comorbid cancer and depression living in rural, low-income communities. Primary hypotheses are that patients randomized to the stepped collaborative care intervention will report clinically meaningful (0.40 or greater effect size) improvements in depression and Quality of Life (QoL) at 6- and 12-months when compared to patients randomized to the screening and referral arm. The secondary hypotheses are that patients randomized to the stepped collaborative care intervention will report clinically meaningful (0.30 or greater effect size) improvements in sleep quality, perceived stress, and social support when compared to the screening and referral arm. The expectation is that caregivers of patients randomized to the intervention arm will have reductions in stress and depression when compared to caregivers of patients randomized to the screening and referral arm. Further exploration will be done of the beneficial effects of the stepped collaborative care intervention on survival.

(Aim 3): To examine the cost-effectiveness of the stepped collaborative care intervention for 242 patients diagnosed with cancer and depression. The stepped collaborative care intervention is expected to be cost-effective compared to the screening and referral arm from the health system perspective in terms of cost per quality-adjusted life year based on established benchmarks for cost-effectiveness. Given the low cost of the intervention and our preliminary data showing reductions in complications and healthcare utilization, there is a high chance that the intervention is, on average, cost saving.

(Aim 4): Guided by the Consolidated Framework for Implementation Science (CFIR), The acceptability, feasibility and actionable factors within the rural context that influence the delivery of the stepped collaborative care intervention will be assessed.. Using mixed methods, guided by the CFIR framework, Surveys will be administered and qualitative interviews performed with patients, caregivers, providers, clinical and research staff after testing the screening and adapted intervention to further refine and inform future implementation in rural, low-income communities.

In terms of relevant prior knowledge and gaps in current knowledge, over 60 million people live in rural communities in the United States. Those who develop cancer are diagnosed later, at more advanced stages, with greater physical comorbidities, poorer quality of life (QoL), and have fewer options for treatment and resources to cope with a diagnosis of cancer when compared to those living in urban communities. As a result, they suffer from greater cancer-related distress and depression. Patients diagnosed with cancer from rural Appalachia were more likely to meet the criteria for clinical levels of distress compared to 27.4% of non-rural cancer patients. Investigators have also observed higher rates of depression in patients from rural, low-income areas when compared to their urban counterparts in Appalachia. Despite the high rates of depression, people who live in rural communities are 47% less likely to receive mental health treatment and 72% less likely to receive specialized mental health treatment when compared to those living in urban communities. Depression results in poorer QoL, decreased adherence to cancer treatments, and increased risk of mortality. Pharmacological and non-pharmacological treatments that have been effective in people from urban communities have not been effective in those living in rural, low-income communities. A stepped collaborative care intervention was designed and tested for socioeconomically disadvantaged patients with comorbid cancer and depression. While the intervention was effective for patients from urban, low-income communities, subgroup analyses revealed the intervention was not effective in patients from rural, low-income communities. While preliminary, there is the belief that cognitive-behavioral therapy (CBT) may not be culturally sensitive in rural, low-income patients. In addition, predictors of depression for these patients included poor sleep, high levels of perceived stress, and lack of social support. The proposal is to adapt the intervention using problem solving therapy, rather than CBT; provide resources to reduce financial stress; and incorporate stress management, support groups, and treatment of sleep problems in the novel intervention. In effort to reduce rural-urban disparities and improve the quality of cancer care, the objectives of this study will be to: (1) adapt the stepped collaborative care intervention to maximize effectiveness for rural, low-income patients, (2) test the effectiveness of the adapted intervention, and (3) prepare for implementation of the intervention in rural, low-income communities.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* biopsy and/or radiograph proven diagnosis of hepatocellular carcinoma, cholangiocarcinoma, gallbladder carcinoma or breast, ovarian, or colorectal cancer with liver metastases with a life expectancy of at least one year;
* age >21 years;
* no evidence of thought disorder, delusions, or active suicidal ideation is observed or reported.

Caregivers:

* a spouse or cohabitating intimate partner of an advanced cancer patient being evaluated at the UPMC's Liver Cancer Center; and
* age >21 years

Exclusion Criteria:

Patients:

* age < 21 years,
* lack of fluency in English,
* evidence of thought disorder, delusions, hallucinations, or suicidal ideation.

Caregivers:

* lack of fluency in English; and
* evidence of thought disorder, delusions, hallucinations, or suicidal ideation.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D)F | Change from baseline in depression at 6 months
  Measure of depression questionnaire- The score is the sum of the 20 questions. Possible range is 0-60. A score of 16 points or more is considered depressed.
Center for Epidemiologic Studies Depression Scale (CES-D) | Change from baseline in depression at 12 months
  Measure of depression questionnaire - The score is the sum of the 20 questions. Possible range is 0-60. A score of 16 points or more is considered depressed.
EuroQOL-5 Dimension Questionnaire (EQ-5D) | Change from baseline in quality of life at 6 months
  Measure of quality of life questionnaire - scale is numbered from 0 to 100. 100 means the best health the participant can imagine. 0 means the worst health the participant can imagine.
EuroQOL-5 Dimension Questionnaire (EQ-5D) | Change from baseline in quality of life at 12 months
  Measure of quality of life questionnaire - scale is numbered from 0 to 100. 100 means the best health the participant can imagine. 0 means the worst health the participant can imagine.

SECONDARY OUTCOMES:
Interpersonal Support Evaluation List (ISEL) | Change from baseline of interpersonal support evaluation at 6 months
  A 12-item measure of perceptions for three dimensions of perceived social support.(Appraisal Support, Belonging Support, Tangible Support) Each dimension is measured by 4 items on a 4-point scale ranging from "Definitely True" to "Definitely False".
Interpersonal Support Evaluation List (ISEL) | Change from baseline of interpersonal support evaluation at 12 months
  A 12-item measure of perceptions for three dimensions of perceived social support.(Appraisal Support, Belonging Support, Tangible Support) Each dimension is measured by 4 items on a 4-point scale ranging from "Definitely True" to "Definitely False".
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline in improved sleep latency at 6 months.
  A measure of sleep quality where respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline in improved sleep latency at 12 months.
  A measure of sleep quality where respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Perceived Stress Scale (PSS) | Change from baseline in perceived stress at 6 months
  This questionnaire about stress is comprised of 14 items intended to measure how unpredictable, uncontrollable, and overloaded individuals find their life circumstances. Individuals rate items on a 5-point Likert scale, ranging from 0 - "Never" to 4 - "Very often." Scores range from 0-56, with higher scores indicating greater perceived stress.
Perceived Stress Scale (PSS) | Change from baseline in perceived stress at 12 months
  This questionnaire about stress is comprised of 14 items intended to measure how unpredictable, uncontrollable, and overloaded individuals find their life circumstances. Individuals rate items on a 5-point Likert scale, ranging from 0 - "Never" to 4 - "Very often." Scores range from 0-56, with higher scores indicating greater perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Steel, PhD, Principal Investigator — UPMC Department of Surgery
Locations (1):
- University of Pittsburgh Medical Centers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analyses plan and all de-identified data collected during the trial may be shared with appropriately credentialed investigators who request data directly from the Primary Investigator:
  Jennifer Steel, PhD, University of Pittsburgh Physicians Department of Surgery Kaufmann Medical Building, Suite 601 3471 Fifth Ave. Pittsburgh, PA 15213 412-692-2041 steejl@upmc.edu.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified data will become available at the end of the study for up to one year following study completion.
Access Criteria: Appropriate investigator credentials (MD, PhD) and direct request for up to one year following study completion